CLINICAL TRIAL: NCT05393427
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of BL-B01D1 in Patients With Locally Advanced or Metastatic Urological Tumors and Other Solid Tumors
Brief Title: A Study of BL-B01D1 in Patients With Locally Advanced or Metastatic Urological Tumors and Other Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: SystImmune Inc. (Industry); Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-102
Record Dates: First submitted 2022-02-20; First posted 2022-05-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced or Metastatic Urinary Tumors; Other Solid Tumors
Keywords: Renal Carcinoma (RCC); Bladder Cancer (BC); Urothelial Cancer (UC); Other Solid Tumors
MeSH Terms: conditions — Carcinoma, Renal Cell; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive BL-B01D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507

SUMMARY:
In phase Ia study, the safety and tolerability of BL-B01D1 in patients with locally advanced or metastatic urinary tumors and other solid tumors will be investigated to determine the dose-limiting toxicity (DLT), maximum tolerated dose (MTD) of BL-B01D1.

In phase Ib study, the safety and tolerability of BL-B01D1 at the phase Ia recommended dose will be further investigated, and recommended phase II dose (RP2D) for phase II clinical studies will be determined.

In addition, the preliminary efficacy, pharmacokinetic characteristics, and immunogenicity of BL-B01D1 in patients with locally advanced or metastatic urinary tumors and other solid tumors will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must sign the informed consent form voluntarily and follow the plan requirements;
2. No gender limit;
3. Age: ≥18 years old and ≤75 years old (stage Ia); ≥18 years old (stage Ib);
4. Expected survival time ≥ 3 months;
5. Locally advanced or metastatic tumors of the urinary system and other solid tumors confirmed by histopathology and/or cytology, which are incurable or currently without standard treatment. Intolerance refers to the occurrence of grade 3-4 adverse reactions after a patient has received standard treatment, and the patient refuses to continue the original treatment;
6. Agree to provide archived tumor tissue specimens (10 unstained sections (anti-extraction) surgical specimens (thickness 4-5μm)) or fresh tissue samples from primary or metastatic lesions within 3 years. If patients cannot provide such specimens, they can be included in the group after the judgment of the investigator if other inclusion criteria are met;
7. Participants must have at least one measurable lesion that meets the definition of RECIST v1.1;
8. Physical fitness score ECOG 0 or 1 point;
9. The toxicity of previous antitumor therapy was restored to ≤ class 1 as defined by NCI-CTCAE v5.0 (the investigators considered asymptomatic laboratory abnormalities such as elevated ALP, hyperuricemia, elevated blood glucose, etc., and toxicities that the investigators judged to be of no safety risk, except for alopecia and grade 2 peripheral neurotoxicity);
10. No serious cardiac dysfunction, left ventricular ejection fraction (LVEF) ≥50%;
11. The organ function must meet the following requirements and standards: a) Bone marrow function: absolute neutrophil count (ANC) ≥1.5×109/L, platelet count ≥75×109/L, hemoglobin ≥90 g/L; B) Liver function: total bilirubin (TBIL≤1.5 ULN), AST and ALT ≤2.5 ULN for participants without liver metastasis, AST and ALT ≤5.0 ULN for liver metastases; c) Kidney function: creatinine (Cr) ≤1.5 ULN, or creatinine clearance (Ccr) ≥50 mL/min (according to the Cockcroft and Gault formula);
12. Coagulation function: International normalized ratio (INR)≤1.5×ULN, and activated partial thromboplastin time (APTT)≤1.5ULN;
13. For premenopausal women with childbearing potential, a pregnancy test must be taken within 7 days prior to the start of treatment. Serum or urine pregnancy must be negative and must be non-lactating; all participants (regardless of male or female) in the group should be treated throughout the treatment. Adequate barrier contraceptive measures should be taken during the treatment and 6 months after the treatment.

Exclusion Criteria:

1. Chemotherapy, biological therapy, immunotherapy, radical radiotherapy, major surgery, targeted therapy (including small molecule inhibitor of tyrosine kinase), and other anti-tumor therapy within 4 weeks or 5 half-lives (whichever is shorter) prior to the first administration; mitomycin and nitrosoureas treatment within 6 weeks prior to the first administration; oral fluorouracil-like drugs such as S-1, capecitabine, or palliative radiotherapy within 2weeks prior to the first administration;
2. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

   1. Have serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias and ⅲ degree ATrioventricular block requiring clinical intervention;
   2. QT interval was prolonged in resting state (QTc > 450 msec for men or 470 msec for women);
   3. Myocardial infarction, unstable angina, cardiac angioplasty or stent implantation, coronary artery/peripheral artery bypass graft, Class ⅲ or ⅳ congestive heart failure, cerebrovascular accident, or transient ischemic attack within 6 months prior to the first administration;
3. Active autoimmune diseases and inflammatory diseases, such as: systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory bowel disease and Hashimoto's thyroiditis, etc., except for type I diabetes, hypothyroidism that can be controlled only by alternative treatment, and skin diseases that do not require systemic treatment (such as vitiligo, psoriasis);
4. Other malignant tumors were diagnosed within 2 years prior to the first administration with the following exceptions: basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or carcinoma in situ after radical resection;
5. Participants have grade 3 lung disease defined according to NCI-CTCAE v5.0, or a history of interstitial lung disease (ILD);
6. Screening for unstable deep vein thrombosis, arterial thrombosis, and pulmonary thrombus requiring therapeutic intervention within the first 6 months Thrombotic events such as stoppage; Thrombus formation associated with infusion set is excluded;
7. Symptoms of active central nervous system metastasis. However, patients with stable brain parenchymal metastases can be enrolled. stable Was defined as: a. duration > 3 months without seizure with or without antiepileptic drugs; b. Have central nervous system (CNS) metastatic and/or cancerous meningitis. He was treated for brain metastases Patients with stable disease for at least 3 months underwent imaging within 28 days before first receiving the study drug Examination determined that no disease progression had occurred and that all neurological symptoms had returned to ≤ grade 1 (CTCAE5.0) Or at baseline (other than signs or symptoms associated with CNS treatment) for at least 2 weeks with no evidence of occurrence Had new or expanded brain metastases and was treated with prednisone within 7 days before first receiving the study drug Patients with dose ≤20mg/ day (or equivalent) were included in this study. Cancer meningitis, regardless of clinical Whether the condition is stable or not should be ruled out;
8. Allergic history to recombinant humanized antibody or mouse chimeric antibody or BL-B01D1 excipients A sensitive patient;
9. Previous recipients of organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
10. The cumulative dose of anthracyclines in previous adjuvant therapy was greater than 360 mg/m2;
11. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus Infection (HBV-DNA copy number > 103 IU/ml) or active hepatitis C virus infection (HCV anti Body positive and HCV-RNA > lower limit of detection);
12. Active infections requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.;
13. The other conditions of participation in this clinical trial were not considered appropriate by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to 21 days after the first dose
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ia: Maximum tolerated dose (MTD) | Up to 21 days after the first dose
  MTD is defined as the highest dose level at which no more than 1 in 6 participants experienced a DLT during the first cycle.
Phase Ib: Recommended Phase II Dose (RP2D) | Up to 21 days after the first dose
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-B01D1

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1 . The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1 .
Cmax | Up to 21 days after the first dose
  Maximum serum concentration (Cmax) of BL-B01D1 will be investigated.
Tmax | Up to 21 days after the first dose
  Time to maximum serum concentration (Tmax) of BL-B01D1 will be investigated.
T1/2 | Up to 21 days after the first dose
  Half-life (T1/2) of BL-B01D1 will be investigated.
AUC0-t | Up to 21 days after the first dose
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
CL (Clearance) | Up to 21 days after the first dose
  CL in the serum of BL-B01D1 per unit of time will be investigated.
Ctrough | Up to 21 days after the first dose
  Ctough is defined as the lowest serum concentration of BL-B01D1 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Incidence and titer of ADA of BL-B01D1 will be evaluated.
Nab (neutralizing antibody) | Up to approximately 24 months
  Incidence and titer of Nab of BL-B01D1 will be evaluated.
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Progression-free Survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-B01D1 to the first date of either disease progression or death, whichever occurs first.
Overall Survival (OS) | Up to approximately 24 months
  The OS is defined as the time from randomization to death (from any cause).

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, PHD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (4):
- China (4):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan